CLINICAL TRIAL: NCT04868604
Title: A Phase I/IIa Theranostic Study of 64Cu-SAR-bisPSMA and 67Cu-SAR-bisPSMA for Identification and Treatment of PSMA-expressing Metastatic Castrate Resistant Prostate Cancer
Brief Title: 64Cu-SAR-bisPSMA and 67Cu-SAR-bisPSMA for Identification and Treatment of PSMA-expressing Metastatic Castrate Resistant Prostate Cancer (SECuRE)
Acronym: SECuRE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP05
Record Dates: First submitted 2021-04-15; First posted 2021-05-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Intervention Model Description: This study is to be conducted in 3 phases, a dosimetry phase, a dose escalation phase and a cohort expansion phase.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 67Cu-SAR-bisPSMA (Experimental): In the dosimetry phase patients will receive a single 200 MBq administration of 64Cu-SAR-bisPSMA.
  In the dose escalation phase patients will receive up to 2 administrations of 200 MBq of 64Cu-SAR-bisPSMA.
  In the cohort expansion phase patients will receive up to 3 administrations of 200 MBq of 64Cu-SAR-bisPSMA.
  In the dose escalation phase patients will receive up to 4 administrations of 67Cu-SAR-bisPSMA (dose will be determined based on cohort allocation).
  In the cohort expansion phase patients will receive up to 6 administrations of 67Cu-SAR-bisPSMA at the recommended dose level determined through dose escalation.
  Interventions: Drug: 64Cu-SAR-bisPSMA; Drug: 67Cu-SAR-bisPSMA

INTERVENTIONS:
Drug: 64Cu-SAR-bisPSMA — 64Cu-SAR-bisPSMA
Drug: 67Cu-SAR-bisPSMA — 67Cu-SAR-bisPSMA

SUMMARY:
The aim of this study is to determine the safety and efficacy of 67Cu-SAR-bisPSMA in participants with PSMA-expressing metastatic castrate resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* ≥18 years of age;
* Eastern Cooperative Oncology Group performance status of 0 to 2;
* Life expectancy >6 months;
* Histological, pathological, and/or cytological confirmation of Prostate cancer (PCa);
* Positive 64Cu-SAR-bisPSMA PET/CT scan, where 64Cu-SAR-bisPSMA uptake (standardized uptake value [SUV] max) of at least 1 known lesion is higher than that of the liver on the 1 hour positron emission tomography (PET)/computed tomography (CT) scan;
* Castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L);
* Have progressive metastatic castration-resistant prostate cancer (mCRPC) despite prior androgen deprivation therapy and:

  * Dose Escalation: at least either enzalutamide and/or abiraterone (or other such androgen receptor pathway inhibitors [androgen receptor pathway inhibitorsARPIs]).
  * Cohort Expansion Main Group: Participant has progressed once or twice on a prior second generation ARPI (abiraterone, enzalutamide, darolutamide, or apalutamide). No concomitant ARPI on study. Note: First generation ARPI is allowed but not considered as prior ARPI. Second generation ARPI must be the most recent therapy received.
  * Cohort Expansion Concomitant Enzalutamide Group: Participant has progressed only once on prior second generation ARPI (prior abiraterone, darolutamide, or apalutamide is allowed, prior treatment with enzalutamide is not allowed). Note: First generation ARPI is allowed but not considered as prior ARPI. Second generation ARPI must be the most recent therapy received.

Documented progressive mCRPC will be based on at least 1 of the following criteria:

1. Serum/plasma prostate specific antigen (PSA) progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimal value for study enrollment is 2.0 ng/mL;
2. Soft-tissue progression defined as a ≥20% increase in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since the last treatment directed at the metastatic cancer has started (not including hormonal therapy) or the appearance of 1 or more new lesions;
3. Progression of bone disease: evaluable disease or new bone lesions(s) by bone scan.

   * ≥1 metastatic lesion that is present at screening CT, magnetic resonance imaging (MRI), or bone scan imaging obtained ≤28 days prior to enrollment into the study;
   * Participants must have recovered to ≤ Grade 2 from all clinically significant toxicities related to prior therapies (prior chemotherapy, radiation, immunotherapy, etc.);
   * Participants must have adequate organ function:

     * Bone marrow reserve:

       * White blood cell (WBC) count ≥2.5 x 109/L (2.5 x 109/L is equivalent to 2.5 x 103/μL and 2.5 x K/μL and 2.5 x 103/cc and 2500/μL) OR
       * Absolute neutrophil count (ANC) ≥1.5 x 109 /L (1.5 x 109 /L is equivalent to 1.5 x 103 /μL and 1.5 x K/μL and 1.5 x 103 /cc and 1500/μL);
     * Platelets ≥100 x 109 /L (100 x 109 /L is equivalent to 100 x 103 /μL and 100 x K/μL and 100 x 103 /cc and 100,000/μL);
     * Hemoglobin ≥9 g/dL (5.59 mmol/L);
     * Total bilirubin ≤1.5 x the institutional upper limit of normal (ULN). For participants with known Gilbert's Syndrome ≤3 x ULN is permitted;
     * Alanine aminotransferase or aspartate aminotransferase ≤3.0 x ULN OR ≤5.0 x ULN for participants with liver metastases;
     * Creatinine clearance or estimated glomerular filtration rate ≥50 mL/min
   * For participants who are human immunodeficiency virus infected: Participant must be healthy and have a low risk of Acquired Immune Deficiency Syndrome related outcomes in the opinion of the Investigator;
   * For participants who have partners of childbearing potential: Partner and/or participant must use a method of birth control with adequate barrier protection.

Exclusion Criteria:

* Major surgery within 12 weeks prior to enrollment into the study;
* Brain metastasis;
* Histologic diagnosis of small cell or neuroendocrine prostate cancer;
* Prior history of leukemia or Myelodysplastic Syndrome;
* Diagnosis of Deep Vein Thrombosis or Pulmonary Embolism within 4 weeks prior to enrollment into the study;
* Unmanageable urinary tract obstruction;
* Evidence of progressive lesion(s) on MRI and/or CT (according to Response Evaluation Criteria in Solid Tumors V1.1) that is prostate-specific membrane antigen (PSMA) negative on the 1 hour 64Cu-SAR-bisPSMA PET/CT scan as determined at screening. NOTE: THIS CRITERION IS NOT APPLICABLE TO PARTICIPANTS IN THE 64Cu-SAR-bisPSMA DOSIMETRY PHASE AND DOSE ESCALATION PHASE.
* Previous treatment with a systemic radionuclide:

  * Dose Escalation: Previous treatment with a systemic radionuclide, including 177Lu, Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Actinium-225, Iodine-131 within 6 months or in case of Radium-223 within 3 months of treatment initiation (Day 0) without prior approval of the medical monitor;
  * Cohort Expansion: Previous treatment with a systemic radionuclide, including Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Iodine-131 within 6 months or in case of Radium-223 within 3 months of treatment initiation (Day 0) without prior approval of the medical monitor; Any previous PSMA targeted radionuclide therapy (including 177Lu and Actinium-225) is also excluded.
* Previous treatment with any systemic anti-cancer therapy (e.g. immunotherapy or biological therapy [including monoclonal antibodies]) within 4 weeks prior to treatment on study with the exception of Luteinizing Hormone Releasing Hormone (LHRH), any other androgen deprivation therapy (ADT) or low dose corticosteroids.

  * Dose Escalation: prior treatment with chemotherapy within 4 weeks of first administration of 67Cu-SAR-bisPSMA is also excluded.
  * Cohort Expansion: Prior treatment with cytotoxic chemotherapy for castration resistant PCa (e.g. taxanes, platinum, estramustine, vincristine, methotrexate, etc) is also excluded. Note: Taxane exposure (maximum 6 cycles) in the adjuvant or neoadjuvant setting is allowed if 12 months have elapsed since completion of this adjuvant or neoadjuvant therapy. Prior treatment with any poly (adenosine diphosphate-ribose) polymerase inhibitors (PARPi) is also excluded. NOTE: THIS CRITERION IS NOT APPLICABLE TO PARTICIPANTS IN THE 64Cu-SAR-bisPSMA DOSIMETRY PHASE;
* Previous treatment with any investigational agents within 4 weeks prior enrollment into the study;
* Known hypersensitivity to the components of the investigational products or its analogues;
* Transfusion for the sole purpose of making a participant eligible for study inclusion;
* Spinal metastasis with symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression;
* Concurrent serious medical conditions, including, but not limited to, New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, known active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation;
* Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, participants with a prior history of malignancy that has been adequately treated and who have been disease free for more than 3 years are eligible, as are participants with adequately treated non-melanoma skin cancer, superficial bladder cancer;
* Any condition or personal situation that would pose an unacceptable radiation safety risk (as per institution guidelines, state and/or national regulations) to the participant or carer at the time of release following the completion of therapy (e.g. uncontrolled urinary incontinence, high dependency care);
* Participants in whom it is known that external beam radiation therapy is scheduled after enrollment into the study. NOTE: THIS CRITERION IS NOT APPLICABLE TO PARTICIPANTS IN THE 64Cu-SAR-bisPSMA DOSIMETRY PHASE.
* Participants in the Cohort Expansion Concomitant Enzalutamide Group:

  1. Participants with known hypersensitivity to enzalutamide or any of its ingredients.
  2. Participants with a history of seizures.
  3. Participants with a history of loss of consciousness (unless of cardiac origin) or transient ischemic attack within 12 months prior to enrolment into the study.
  4. Participants with conditions that increase the risk of seizures include those with a history of traumatic brain injury, stroke or cerebrovascular disease, arteriovenous malformations in the brain, neurodegenerative diseases, primary or metastatic brain tumors, active leptomeningeal disease, uncontrolled hypertension (systolic >179 or diastolic >105), patients undergoing alcohol withdrawal.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of 64Cu-SAR-bisPSMA | 48 hours
  Biodistribution will be calculated by utilizing the PET/CT scans.
Dosimetry of 64Cu-SAR-bisPSMA | 48 hours
  Dosimetry will be calculated by utilizing the PET/CT scans.
Modelling of 67Cu-SAR-bisPSMA dosimetry utilizing the 64Cu-SAR-bisPSMA PET/CT scans | 48 hours
  Dosimetry will be calculated by utilizing the PET/CT scans.
Maximum Tolerated Dose (MTD) or Maximum Feasible Dose of a single dose of 67Cu-SAR-bisPSMA | 8 weeks
  MDT as determined by cohort observations of dose limiting toxicities (DLT)
Recommended dose of two doses of 67Cu-SAR-bisPSMA | 14 weeks
  Recommended dose as determined by cohort observations of DLTs
Efficacy of 67Cu-SAR-bisPSMA in terms of Prostate specific Antigen (PSA) response | Up to 5 years
  Proportion of participants with ≥50% decline in PSA
Efficacy of 67Cu-SAR-bisPSMA in terms of radiographic response | Up to 5 years
  Efficacy will be assessed via the overall response rate according to RECIST V1.1 for soft tissue disease and according PCWG3 for bone lesions
Incidence of 67Cu-SAR-bisPSMA Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 5 years
  Adverse Events will be as assessed by CTCAE version 5.00
Safety and tolerability of 67Cu-SAR-bisPSMA: Number of Participants With Changes from baseline in Vital Signs | Up to 1 year
  Change from baseline in vital signs
Safety and tolerability of 67Cu-SAR-bisPSMA: Number of Participants With Changes from baseline in electrocardiogram (ECG) parameters | Up to 24 weeks
  Change from baseline in ECG parameters
Safety and tolerability of 67Cu-SAR-bisPSMA: Number of Participants With Changes from baseline in laboratory results | Up to 22 weeks
  Change from baseline in laboratory results
Incidence of 64Cu-SAR-bisPSMA Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 5 years
  Adverse Events will be as assessed by CTCAE version 5.00

CONTACTS AND LOCATIONS:
Overall Officials: Clarity Pharmaceuticals, Study Director — Clarity Pharmaceuticals
Locations (7):
- United States (7):
  - Stanford Cancer Institute, Stanford, California
  - East Jefferson General Hospital, River Ridge, Louisiana
  - BAMF Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine at Barnes-Jewish Hospital, St Louis, Missouri
  - XCancer, Omaha, Nebraska
  - Weill Cornell Medicine at New York-Presbyterian, New York, New York